CLINICAL TRIAL: NCT01190475
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled Study of Oral BGS649 Monotherapy Assessing Safety and Tolerability in Patients With Moderate to Severe Endometriosis
Brief Title: BGS649 Monotherapy in Moderate to Severe Endometriosis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mereo BioPharma (Industry)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CBGS649A2105
Record Dates: First submitted 2010-08-19; First posted 2010-08-27 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-10

CONDITIONS: Endometriosis
Keywords: Endometriosis; Infertility; Pain; Vaginal Diseases; Uterine Diseases
MeSH Terms: conditions — Endometriosis; Infertility; Pain; Vaginal Diseases; Uterine Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- BGS649 high dose (Experimental): 1 BGS649 1.0mg capsule with three 0.1 mg placebo capsules.
  Interventions: Drug: Active treatment with a high dose of BGS649
- BGS649 low dose (Experimental): 1 BGS649 1.0 mg placebo capsule and 3 BGS649 0.1 mg capsules
  Interventions: Drug: Active treatment with a low dose of BGS649
- Placebo to BGS649 (Placebo Comparator): 1 matching placebo 1.0mg matching and three matching 0.1 mg placebo capsules
  Interventions: Drug: Placebo treatment to blind study

INTERVENTIONS:
Drug: Active treatment with a high dose of BGS649
  Arms: BGS649 high dose
Drug: Active treatment with a low dose of BGS649
  Arms: BGS649 low dose
Drug: Placebo treatment to blind study
  Arms: Placebo to BGS649

SUMMARY:
This study will assess the safety and tolerability of BGS649 in women with moderate to severe endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women with documented moderate to severe endometriosis. Occurrence of three sequential menstrual cycles of 24-35 days duration prior to enrollment.
* Laparoscopically proven diagnosis of moderate to severe endometriosis (diagnosed within the past 10 years before screening).
* Patients not planning to become pregnant within one year after the screening visit and willing to use two effective methods of non-hormonal, barrier birth control for the duration of the study or who are surgically sterile.
* Patients must have a score of at least 4 on the numerical rating scale (NRS) for one of the following three pain measurements: pelvic pain, menstrual pain and dyspareunia

Exclusion Criteria:

* Estrogen replacement therapy using either prescription medications or estrogen-containing OTC nutritional/herbal supplements such as soy extracts or topical estrogens.
* Aromatase inhibitor therapy (includes Femara (letrozole), Aromasin (exemestane) or Arimidex (anastrozole) within the past 12 months.
* Oral bisphosphonate therapy (i.e. Fosamax (alendronate)) within the past 6 months or intravenous bisphosphonate (i.e., Reclast, pamidronate) < 15 months from screening.
* Systemic glucocorticoid therapy within the past 4 weeks.
* Contra-indications to oral contraceptive use.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Parkin, PhD FRCP, Study Director — Mereo BioPharma
Locations (1):
- Novartis Investigative Site, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: 1 matching placebo 1.0mg matching and three matching 0.1 mg placebo capsules
Period: Overall Study
Arm/Group | BGS649 High Dose | BGS649 Low Dose | Placebo
Started | 2 | 2 | 2
Completed | 2 | 2 | 1
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BGS649 High Dose | BGS649 Low Dose | Placebo | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 30 [21 to 39] | 28 [28 to 28] | 30.5 [30 to 31] | 29 [21 to 39]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 6
  Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 1 | 2 | 2 | 5
  Black | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Develop 2 or More Follicles With Diameter 16 mm or Larger
Description: Proportion of patients who develop 2 or more follicles with diameter 16 mm or larger.
Time Frame: 8 months
Population: Proportion of patients who develop 2 or more follicles with diameter 16 mm or larger
Measure: Count of Participants; unit: Participants
Groups:
- BGS649 High Dose; BGS649 Low Dose: BGS649
- Placebo: Placebo
Arm/Group | BGS649 High Dose | BGS649 Low Dose | Placebo
Number analyzed (Participants) | 2 | 2 | 2
Participants | 2 | 2 | 0

2. Secondary Outcome: Pharmacokinetic Profille of BGS649 as Described by AUC0-672h
Description: AUC0-672 is a measurement of how much drug reaches a person's bloodstream in a given period of time after a dose is given. Measurements were performed at dose 1 (in cycle 2) and after dose 2 (in cycle 4). Sampling occured at pre-dose, 0.5-1.5h and 4-8 h post-dose.
Time Frame: 8 hours
Population: Full analysis set
Measure: Mean (Full Range); unit: ng*hr/mL
Groups:
- BGS649 High Dose: 1 BGS649 1.0mg capsule with three 0.1 mg placebo capsules.
  Active treatment with a high dose of BGS649
- BGS649 Low Dose: 1 BGS649 1.0 mg placebo capsule and 3 BGS649 0.1 mg capsules
  Active treatment with a low dose of BGS649
Arm/Group | BGS649 High Dose | BGS649 Low Dose
Number analyzed (Participants) | 2 | 2
ng*hr/mL
  AUC0-672 at Cycle 2 | 2557 [2430 to 2690] | 443.8 [443.8 to 443.8]
  AUC0-672 at Cycle 4 | 3283 [2960 to 3610] | 639.6 [639.6 to 639.6]

3. Secondary Outcome: Pharmacokinetic Profile of BGS649 as Described by Cmax
Description: The peak plasma concentration of BGS649 after dosing at cycle 2 and cycle 4. Measurements were performed at dose 1 (in cycle 2) and after dose 2 (in cycle 4). Sampling occured at pre-dose, 0.5-1.5h and 4-8 h post-dose.
Time Frame: 8 hours
Population: Pharmacokinetic patient population. Study met the pre-defined safety stopping criteria and so was not fully enrolled. The PK results of for one of the patients could not be reported - missing data for cycle 2 and meeting the stopping criteria before cycle 4.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | BGS649 High Dose | BGS649 Low Dose
Number analyzed (Participants) | 2 | 1
ng/mL
  Cycle 2 | 9.040 (4.0447) | 2.720
  Cycle 4 | 15.25 (0.91924) | 3.410

4. Secondary Outcome: Pharmacokinetic Profile of BGS649 as Described by Tmax
Description: Time taken to reach the maximum concentration in plasma of BGS649 at cycle 2 and cycle 4. Measurements were performed at dose 1 (in cycle 2) and after dose 2 (in cycle 4). Sampling occurred at pre-dose, 0.5-1.5h and 4-8 h post-dose.
Time Frame: 8 hours
Population: as for outcome 3
Measure: Mean (Full Range); unit: hours
Arm/Group | BGS649 High Dose | BGS649 Low Dose
Number analyzed (Participants) | 2 | 1
hours
  Cycle 2 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  Cycle 4 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]

ADVERSE EVENTS:
Arm/Group | BGS649 High Dose | BGS649 Low Dose | Placebo
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BGS649 High Dose (N=2) | BGS649 Low Dose (N=2) | Placebo (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was prematurely terminated because the safety endpoint was reached after a total of 6 patients were randomized into one of the 3 treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All PIs must seek written permission from the sponsor prior to publication of any trial results.